CLINICAL TRIAL: NCT05018104
Title: Development and Internal Validation of a Multivariable Risk Prediction Model for Severe Rebound Pain After Lower Limb Orthopedic Surgery Involving Single-Shot Popliteal Sciatic Nerve Blocks: A Single Centre Retrospective Cohort Study
Brief Title: Risk Model for Severe Rebound Pain After Lower Limb Orthopedic Surgery Involving Single-Shot Sciatic Nerve Blocks
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Cynthia Yarnold, Clinical Assistant Professor, University of British Columbia
Other Study IDs: H20-01349
Record Dates: First submitted 2021-08-10; First posted 2021-08-24 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Orthopedic Procedures; Pain, Postoperative; Surgery; Nerve Block; Ambulatory Surgical Procedures; Pain
Keywords: Rebound Pain; Continous Popliteal Sciatic Nerve Block Catheter; Orthopedic Surgery
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lower Limb Orthopedic Surgery Patients who Received Popliteal Sciatic Nerve Blocks: All patients undergoing lower limb surgery who received popliteal sciatic nerve blocks (with or without other peripheral nerve blocks) at St. Paul's Hospital from January 4, 2016 to November 1, 2019
  Interventions: Other: This is not an interventional study

INTERVENTIONS:
Other: This is not an interventional study — This study utilizes data from the St. Paul's Hospital Peripheral Nerve Block Database.

SUMMARY:
Rebound pain is a well-recognized phenomenon after the effects of a nerve block wear off. Severe rebound pain can happen after outpatient surgery, with patients often needing to come back to the hospital or use other health care resources.

People who are younger, female or have more pain before surgery are at higher risk of having rebound pain. Bone surgeries and upper limb surgeries also increase the chances of having rebound pain after surgery. Patients who have a tourniquet used during leg surgery often have worse pain after surgery compared to patients who get surgery without the use of a tourniquet.

Things that may reduce the chances of getting rebound pain are the use of nerve block catheters, certain additives in nerve blocks and using multiple types of pain killers before the block wears off. Using nerve block catheters can be expensive, so a targeted approach of giving these catheters to patients who have the highest chances of getting rebound pain may be the best way to allocate resources and help patients.

The aim of this study is to create and test a risk model for severe rebound pain after lower limb surgery where patients are getting a sciatic nerve block.

DETAILED DESCRIPTION:
Rebound pain is a well-recognized phenomenon after the resolution of peripheral nerve blocks. Severe rebound pain is prevalent after ambulatory surgery, with potential resultant increased health-care utilization and cost. Risk factors for severe rebound pain may include younger age, female sex, high preoperative pain score, bone surgeries, and upper limb surgeries. Use of tourniquet for lower limb procedures is also associated with worse postoperative pain compared to without. Protective factors may include continuous perineural catheter, regional anesthesia adjuncts, and multimodal oral pain management prior to resolution of peripheral nerve blockade. However, placement of continuous peripheral nerve block catheters utilizes additional health care resources; hence, a targeted approach where continuous perineural catheters are offered to patients at the highest risk of severe rebound pain could potentially offer the biggest benefit.

The aim of the study is to derive and validate a multivariable prediction model for severe rebound pain after lower limb surgery involving popliteal blockade, to assist with risk stratification and shared decision making.

The primary model endpoint is severe rebound pain, defined by transition from well-controlled pain (numerical rating scale [NRS] 3 or less or patient report of satisfactory pain control) in the post anesthetic care unit (PACU) while the block is working to severe pain (NRS pain score 7 or greater) within 48 h of block performance. This definition is modified from that of Barry et al., 2020 as clinically, the investigators have noted some patients having sensory blocks lasting more than 24 hours with the use of adjuncts.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent lower limb surgery and received a single-shot popliteal sciatic nerve block pre-operatively at St. Paul's Hospital from January 4, 2016 to November 1, 2019

Exclusion Criteria:

* Patients who had uncontrolled pain (defined as NRS greater than 3 and/or nursing note documentation of uncontrolled or severe pain and/or undocumented pain status) in the post anesthesia care unit (post-operatively)
* Patients who received a popliteal sciatic nerve catheter

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients who received a single-shot popliteal sciatic nerve block at St. Paul's Hospital in the study period.
Sampling Method: Non-Probability Sample
Enrollment: 1270 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
Area Under the Receiver Operating Characteristic (ROC) Curve | Not a time dependent outcome (retrospective participant pain data up to 48 hours after a nerve block was administered)
  The Area under the ROC Curve provides a graphical display of sensitivity and specificity and is used to evaluate the discriminative ability of the risk prediction model.
Calibration Slope | Not a time dependent outcome (model validation test based on retrospective participant pain data up to 48 hours after a nerve block was administered)
  To evaluate the the degree to which numerical predictions are too high or too low compared to outcomes.

SECONDARY OUTCOMES:
Scaled Brier Score | Not a time dependent outcome (model evaluation/validation test based on retrospective participant pain data up to 48 hours after a nerve block was administered)
  A proper score function that measures the accuracy of probabilistic predictions.
Nagelkerke R2 | Not a time dependent outcome (model evaluation/validation test based on retrospective participant pain data up to 48 hours after a nerve block was administered)
  An adjusted version of the Cox & Snell R-square that adjusts the scale of the statistic to cover the full range from 0 to 1.
Decile Calibration Plots | Not a time dependent outcome (model evaluation/validation test based on retrospective participant pain data up to 48 hours after a nerve block was administered)
  Decile Calibration Plots will be generated for the final prediction models to further assess calibration, with Loess-smoothed calibration curves created for each imputed dataset.
Decision Curve Analysis | Not a time dependent outcome (model evaluation/validation test based on retrospective participant pain data up to 48 hours after a nerve block was administered)
  The Decision Curve Analysis is a method to evaluate prediction models and diagnostic tests. It will be performed on the final prediction models.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Yarnold, MD, Principal Investigator — University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jen TTH, Ke JXC, Wing KJ, Denomme J, McIsaac DI, Huang SC, Ree RM, Prabhakar C, Schwarz SKW, Yarnold CH. Development and internal validation of a multivariable risk prediction model for severe rebound pain after foot and ankle surgery involving single-shot popliteal sciatic nerve block. Br J Anaesth. 2022 Jul;129(1):127-135. doi: 10.1016/j.bja.2022.03.030. Epub 2022 May 12. PMID 35568510

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-26): https://cdn.clinicaltrials.gov/large-docs/04/NCT05018104/Prot_SAP_000.pdf